CLINICAL TRIAL: NCT03511820
Title: A Post Marketing Surveillance Study of Lipo-AB® (Amphotericin B) in Neutropenic Patients With Persistent Fever
Status: Completed | Type: Observational
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Other Study IDs: TTYLA1201
Record Dates: First submitted 2018-04-01; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Neutropenia, Febrile
Keywords: Amphotericin B; liposome; post marketing surveillance
MeSH Terms: conditions — Febrile Neutropenia | interventions — Amphotericin B; Liposomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lipo-AB® (amphotericin B) liposome — 1. Name: Lipo-AB® (amphotericin B) liposome for injection
  2. Dosage form: Lyophilized powder 50 mg/vial
  3. Dose: Based on approved package insert and physician's discretion Recommended initial dose: 3 mg/kg/day
  4. Dosing schedule:
  All patients will receive Lipo-AB® based on the approved package insert and physician's clinical decision.

SUMMARY:
Amphotericin B is a polyene antifungal drug used for the treatment of many systemic fungal infections. It is associated with many side effects which in some cases can be very severe and potentially lethal. Lipo-AB® is a true single bilayer liposomal drug delivery system, consisting of unilamellar bilayer liposomes with amphotericin B intercalated within the membrane. Prior studies showed that the liposomal formulation of amphotericin B greatly reduces the side effects of the parent drug, such as nephrotoxicity. This study is designed to evaluate the safety and efficacy of Lipo-AB® in neutropenic patients with persistent fever in routine clinical practice in Taiwan.

1. Primary objective:

   • To evaluate the nephrotoxicity of Lipo-AB® (amphotericin B) treatment in neutropenic patients with persistent fever in Taiwan clinical practice.
2. Secondary objectives:

(1) To evaluate the safety profile of Lipo-AB® (amphotericin B) in neutropenic patients with persistent fever in Taiwan clinical practice.

(2) To evaluate the treatment efficacy of Lipo-AB® (amphotericin B) in neutropenic patients with persistent fever in Taiwan clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male with no age limit
2. Patient for whom Lipo-AB® is medically recommended due to following conditions:

   * Absolute neutrophil count (ANC) < 500/mm3 for at least 96 hours
   * Received parenteral broad spectrum antibacterial therapy for at least 96 hours
   * Fever of ≥ 38.0°C (tympanic temperature)
3. Subject or his/her legally acceptable representative is willing and able to provide a written informed consent

Exclusion Criteria:

1. Pregnant female, with the exception of those for whom the possible benefits to be derived outweigh the potential risks involved
2. Use of other investigational product 2 weeks before the initiation of Lipo-AB® treatment which is considered not suitable for this study by investigator
3. Use of any parenteral antifungals for current infection which is not considered treatment failure (either intolerance to the drug or lack of response)
4. Any condition which is considered not suitable for liposomal amphotericin B therapy by investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neutropenic patients with persistent fever who are recommended to receive systemic antifungal therapy based on physician's decision will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence rate of nephrotoxicity | through Observation period (up to 44 days)
  * Nephrotoxicity is defined as serum creatinine (SCr) values increasing 100% or more over pretreatment levels in pediatric patients, and creatinine values increasing 100% or more over pretreatment levels in adult patients provided the peak creatinine concentration was > 1.2 mg/dL during treatment period.
  ** The nephrotoxicity associated with baseline SCr will also be assessed.

SECONDARY OUTCOMES:
Categorization of the change in renal function | through Observation period (up to 44 days)
  * SCr < 1.5 x baseline SCr (BSC)
  * SCr ≥ 1.5 x BSC
  * SCr ≥ 2 x BSC
  * SCr ≥ 3 x BSC
Change in laboratory parameters (1) | through Observation period (up to 44 days)
  hemoglobin (Hb in g/dL)
Change in laboratory parameters (2) | through Observation period (up to 44 days)
  hematocrit (Hct in %)
Change in laboratory parameters (3) | through Observation period (up to 44 days)
  red blood cell (RBC in 10^6/uL)
Change in laboratory parameters (4) | through Observation period (up to 44 days)
  white blood cell (WBC in 10^3/uL)
Change in laboratory parameters (5) | through Observation period (up to 44 days)
  ANC (absolute neutrophil count in mm^3)
Change in laboratory parameters (6) | through Observation period (up to 44 days)
  platelet count in 10^3/uL
Change in laboratory parameters (7) | through Observation period (up to 44 days)
  alanine aminotransferase (ALT in U/L)
Change in laboratory parameters (8) | through Observation period (up to 44 days)
  aspartate aminotransferase (AST in U/L)
Change in laboratory parameters (9) | through Observation period (up to 44 days)
  total bilirubin (TB in mg/dL)
Change in laboratory parameters (10) | through Observation period (up to 44 days)
  BUN in mg/dL
Change in laboratory parameters (11) | through Observation period (up to 44 days)
  serum creatinine (SCr in mg/dL)
Change in laboratory parameters (12) | through Observation period (up to 44 days)
  glucose (mg/dL)
Change in laboratory parameters (13) | through Observation period (up to 44 days)
  Na (mmol/L)
Change in laboratory parameters (14) | through Observation period (up to 44 days)
  K (mmol/L)
Change in laboratory parameters (15) | through Observation period (up to 44 days)
  Mg (mg/dL)
Change in laboratory parameters (16) | through Observation period (up to 44 days)
  Ca (mg/dL)
Change in laboratory parameters (17) | through Observation period (up to 44 days)
  Urine protein (mg/dL)
Change in vital signs (1) | through Observation period (up to 44 days)
  systolic/diastolic blood pressure (SBP/ DBP in mmHg)
Change in vital signs (2) | through Observation period (up to 44 days)
  pulse rate (PR in bpm)
Change in vital signs (3) | through Observation period (up to 44 days)
  tympanic temperature (TT in °C)
Adverse event(s) | through Observation period (up to 44 days)
  Hypokalemia, Hypomagnesemia, Hypocalcemia, Hypernatremia, Hyponatremia, Infusion-related reaction(s) (IRR), Other adverse event(s).
Overall success rate | through Observation period (up to 44 days)
  Defined as a composite of five criteria:
  * Survival for 7 days after completion of the observational treatment
  * Fever resolved during neutropenic period: defined as a tympanic temperature < 38°C for at least 48 hours
  * Baseline fungal infection cured (if present): defined as (i) resolution of all attributable clinical symptoms and signs of fungal infection during the observational period, (ii) negative microbiological result at the EOT (end of treatment), if available
  * No breakthrough fungal infections (proved, probable and possible) during administration of the observational drug or within 7 days after the completion of observational treatment
  * Absence of premature discontinuation of the observational drug because of toxicity or lack of efficacy
Overall survival rate | through Observation period (up to 44 days)

CONTACTS AND LOCATIONS:
Locations (9):
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Mucinipal Wanfang Hospital, Taipei
  - Chang Guang Memorial Hospital at LinKou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No